CLINICAL TRIAL: NCT03808298
Title: A Single-Center, Multiple-Dose, Randomized, Double-Blind, Placebo-Controlled, Cross-Over Study to Investigate the Effect of Balovaptan on the QTC Interval in Healthy Subjects
Brief Title: Study to Investigate the Effect of Balovaptan on the QTC Interval in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: WP40734
Record Dates: First submitted 2019-01-07; First posted 2019-01-17 (Actual); Results first posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Treatment Sequence 1: A, B, C (Experimental)
  Interventions: Drug: Balovaptan therapeutic dose Treatment A; Drug: Balovaptan supra-therapeutic dose Treatment B; Drug: Active control [moxifloxacin] on Day 2 Treatment C; Drug: Placebo for Balovaptan Treatment C; Drug: Placebo for Moxifloxacin Treatment A; Drug: Placebo for Moxifloxacin Treatment B; Drug: Moxifloxacin Treatment C; Drug: Placebo for Moxifloxacin Treatment C
- Treatment Sequence 2: A, C, B (Experimental)
  Interventions: Drug: Balovaptan therapeutic dose Treatment A; Drug: Balovaptan supra-therapeutic dose Treatment B; Drug: Active control [moxifloxacin] on Day 2 Treatment C; Drug: Placebo for Balovaptan Treatment C; Drug: Placebo for Moxifloxacin Treatment A; Drug: Placebo for Moxifloxacin Treatment B; Drug: Moxifloxacin Treatment C; Drug: Placebo for Moxifloxacin Treatment C
- Treatment Sequence 3: B, A, C (Experimental)
  Interventions: Drug: Balovaptan therapeutic dose Treatment A; Drug: Balovaptan supra-therapeutic dose Treatment B; Drug: Active control [moxifloxacin] on Day 2 Treatment C; Drug: Placebo for Balovaptan Treatment C; Drug: Placebo for Moxifloxacin Treatment A; Drug: Placebo for Moxifloxacin Treatment B; Drug: Moxifloxacin Treatment C; Drug: Placebo for Moxifloxacin Treatment C
- Treatment Sequence 4: B, C, A (Experimental)
  Interventions: Drug: Balovaptan therapeutic dose Treatment A; Drug: Balovaptan supra-therapeutic dose Treatment B; Drug: Active control [moxifloxacin] on Day 2 Treatment C; Drug: Placebo for Balovaptan Treatment C; Drug: Placebo for Moxifloxacin Treatment A; Drug: Placebo for Moxifloxacin Treatment B; Drug: Moxifloxacin Treatment C; Drug: Placebo for Moxifloxacin Treatment C
- Treatment Sequence 5: C, A, B (Experimental)
  Interventions: Drug: Balovaptan therapeutic dose Treatment A; Drug: Balovaptan supra-therapeutic dose Treatment B; Drug: Active control [moxifloxacin] on Day 2 Treatment C; Drug: Placebo for Balovaptan Treatment C; Drug: Placebo for Moxifloxacin Treatment A; Drug: Placebo for Moxifloxacin Treatment B; Drug: Moxifloxacin Treatment C; Drug: Placebo for Moxifloxacin Treatment C
- Treatment Sequence 6: C, B, A (Experimental)
  Interventions: Drug: Balovaptan therapeutic dose Treatment A; Drug: Balovaptan supra-therapeutic dose Treatment B; Drug: Active control [moxifloxacin] on Day 2 Treatment C; Drug: Placebo for Balovaptan Treatment C; Drug: Placebo for Moxifloxacin Treatment A; Drug: Placebo for Moxifloxacin Treatment B; Drug: Moxifloxacin Treatment C; Drug: Placebo for Moxifloxacin Treatment C
- Treatment Sequence 7: A, B, D (Experimental)
  Interventions: Drug: Balovaptan therapeutic dose Treatment A; Drug: Balovaptan supra-therapeutic dose Treatment B; Drug: Active control [Moxifloxacin] on Day 15 Treatment D; Drug: Placebo for Balovaptan Treatment D; Drug: Placebo for Moxifloxacin Treatment A; Drug: Placebo for Moxifloxacin Treatment B; Drug: Placebo for Moxifloxacin Treatment D; Drug: Moxifloxacin Treatment D
- Treatment Sequence 8: A, D, B (Experimental)
  Interventions: Drug: Balovaptan therapeutic dose Treatment A; Drug: Balovaptan supra-therapeutic dose Treatment B; Drug: Active control [Moxifloxacin] on Day 15 Treatment D; Drug: Placebo for Balovaptan Treatment D; Drug: Placebo for Moxifloxacin Treatment A; Drug: Placebo for Moxifloxacin Treatment B; Drug: Placebo for Moxifloxacin Treatment D; Drug: Moxifloxacin Treatment D
- Treatment Sequence 9: B, A, D (Experimental)
  Interventions: Drug: Balovaptan therapeutic dose Treatment A; Drug: Balovaptan supra-therapeutic dose Treatment B; Drug: Active control [Moxifloxacin] on Day 15 Treatment D; Drug: Placebo for Balovaptan Treatment D; Drug: Placebo for Moxifloxacin Treatment A; Drug: Placebo for Moxifloxacin Treatment B; Drug: Placebo for Moxifloxacin Treatment D; Drug: Moxifloxacin Treatment D
- Treatment Sequence 10: B, D, A (Experimental)
  Interventions: Drug: Balovaptan therapeutic dose Treatment A; Drug: Balovaptan supra-therapeutic dose Treatment B; Drug: Active control [Moxifloxacin] on Day 15 Treatment D; Drug: Placebo for Balovaptan Treatment D; Drug: Placebo for Moxifloxacin Treatment A; Drug: Placebo for Moxifloxacin Treatment B; Drug: Placebo for Moxifloxacin Treatment D; Drug: Moxifloxacin Treatment D
- Treatment Sequence 11: D, A, B (Experimental)
  Interventions: Drug: Balovaptan therapeutic dose Treatment A; Drug: Balovaptan supra-therapeutic dose Treatment B; Drug: Active control [Moxifloxacin] on Day 15 Treatment D; Drug: Placebo for Balovaptan Treatment D; Drug: Placebo for Moxifloxacin Treatment A; Drug: Placebo for Moxifloxacin Treatment B; Drug: Placebo for Moxifloxacin Treatment D; Drug: Moxifloxacin Treatment D
- Treatment Sequence 12: D, B, A (Experimental)
  Interventions: Drug: Balovaptan therapeutic dose Treatment A; Drug: Balovaptan supra-therapeutic dose Treatment B; Drug: Active control [Moxifloxacin] on Day 15 Treatment D; Drug: Placebo for Balovaptan Treatment D; Drug: Placebo for Moxifloxacin Treatment A; Drug: Placebo for Moxifloxacin Treatment B; Drug: Placebo for Moxifloxacin Treatment D; Drug: Moxifloxacin Treatment D

INTERVENTIONS:
Drug: Balovaptan therapeutic dose Treatment A — Days 1-14: A single once daily dose at dose level A of balovaptan for 14 days
Drug: Balovaptan supra-therapeutic dose Treatment B — Days 1-14: A single once daily oral dose at dose level B of balovaptan for 14 days.
Drug: Active control [moxifloxacin] on Day 2 Treatment C — Day 2: A single oral dose of 400 mg moxifloxacin capsule.
  Arms: Treatment Sequence 1: A, B, C; Treatment Sequence 2: A, C, B; Treatment Sequence 3: B, A, C; Treatment Sequence 4: B, C, A; Treatment Sequence 5: C, A, B; Treatment Sequence 6: C, B, A
Drug: Active control [Moxifloxacin] on Day 15 Treatment D — Day 15: A single oral dose of 400 mg moxifloxacin capsule.
  Arms: Treatment Sequence 10: B, D, A; Treatment Sequence 11: D, A, B; Treatment Sequence 12: D, B, A; Treatment Sequence 7: A, B, D; Treatment Sequence 8: A, D, B; Treatment Sequence 9: B, A, D
Drug: Placebo for Balovaptan Treatment C — Days 1-14: Matching placebo for balovaptan for 14 days.
  Arms: Treatment Sequence 1: A, B, C; Treatment Sequence 2: A, C, B; Treatment Sequence 3: B, A, C; Treatment Sequence 4: B, C, A; Treatment Sequence 5: C, A, B; Treatment Sequence 6: C, B, A
Drug: Placebo for Balovaptan Treatment D — Days 1-14: Matching placebo for balovaptan for 14 days.
  Arms: Treatment Sequence 10: B, D, A; Treatment Sequence 11: D, A, B; Treatment Sequence 12: D, B, A; Treatment Sequence 7: A, B, D; Treatment Sequence 8: A, D, B; Treatment Sequence 9: B, A, D
Drug: Placebo for Moxifloxacin Treatment A — Day 2 and 15: A single oral dose of a matching placebo capsule for moxifloxacin.
Drug: Placebo for Moxifloxacin Treatment B — Days 2 and 15: Single oral dose of a matching placebo capsule of moxifloxacin.
Drug: Moxifloxacin Treatment C — Day 2: A single oral dose of 400 mg moxifloxacin capsule.
  Arms: Treatment Sequence 1: A, B, C; Treatment Sequence 2: A, C, B; Treatment Sequence 3: B, A, C; Treatment Sequence 4: B, C, A; Treatment Sequence 5: C, A, B; Treatment Sequence 6: C, B, A
Drug: Placebo for Moxifloxacin Treatment C — Day 15: A single oral dose of a matching placebo capsule for moxifloxacin.
  Arms: Treatment Sequence 1: A, B, C; Treatment Sequence 2: A, C, B; Treatment Sequence 3: B, A, C; Treatment Sequence 4: B, C, A; Treatment Sequence 5: C, A, B; Treatment Sequence 6: C, B, A
Drug: Placebo for Moxifloxacin Treatment D — Day 2: A single oral dose of a matching placebo capsule for moxifloxacin.
  Arms: Treatment Sequence 10: B, D, A; Treatment Sequence 11: D, A, B; Treatment Sequence 12: D, B, A; Treatment Sequence 7: A, B, D; Treatment Sequence 8: A, D, B; Treatment Sequence 9: B, A, D
Drug: Moxifloxacin Treatment D — Day 15: A single oral dose of 400 mg moxifloxacin capsule.
  Arms: Treatment Sequence 10: B, D, A; Treatment Sequence 11: D, A, B; Treatment Sequence 12: D, B, A; Treatment Sequence 7: A, B, D; Treatment Sequence 8: A, D, B; Treatment Sequence 9: B, A, D

SUMMARY:
This was a single-center, multiple-dose, randomized, double-blind, placebo-controlled, positive-controlled, twelve sequence, 3-period cross-over study to investigate the effect of balovaptan on the QTc interval in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects. Healthy status is defined by absence of evidence of any active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead ECG, hematology, blood chemistry, urinalysis, and serology.
* Body Mass Index of 18 to 30 kg/m2, inclusive.
* For women of childbearing potential: agreement to use at least 1 acceptable form of contraception during the entire study and for 90 days following last dose of study drug.
* For men: vasectomized, agreement to remain abstinent or use of a condom during intercourse. Must also agree to refrain from donating sperm.
* Fluent in English.

Exclusion Criteria:

* If female, a positive pregnancy test at screening or prior to Day 1 of any Treatment Period.
* Lactating women.
* Any condition or disease detected during the medical interview / physical examination that would render the subject unsuitable for the study, place the subject at undue risk or interfere with the ability of the subject to complete the study in the opinion of the Investigator or designee.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2019-06-14 (Actual); Study Completion 2019-07-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- PRA International Clinical Pharmacology Center (EDS US Clinic), Lenexa, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Sequence A and B and Either C or D: All participants received Treatment A and Treatment B and either Treatment C or Treatment D.
Period: Overall Study
Arm/Group | Treatment Sequence A and B and Either C or D
Started | 57
Completed | 49
Not Completed | 8
Not completed — Adverse Event | 3
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1
Not completed — Positive Urine Drug Screen at Check-in | 3

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Sequence A and B and Either C or D
Number analyzed (Participants) | 57
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.9 (10.59)
Age, Continuous [Median (Full Range); unit: Years] | 36 [18 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 52
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 31
  White | 23
  More than one race | 3
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change-From-Baseline QTcF at Dose Level B Measured on 12-Lead ECGs Extracted From Continuous Recordings
Description: Change-from-baseline QTcF (ΔΔQTcF) at dose level B of balovaptan measured on 12-lead ECGs extracted from continuous recordings at the specified time points on Day 14.
Time Frame: Baseline (Predose Day 1), Day 14. (Each treatment period is 15 days.)
Population: QT/QTc population included all participants in the Safety population with ECG measurements at baseline as well as on treatment with at least 1 post-dose time point with a valid ΔQTcF value.
Measure: Least Squares Mean (90% Confidence Interval); unit: ms
Groups:
- Dose Level B of Balovaptan: Participants received dose level of B balovaptan.
- Placebo: Participants received placebo.
Arm/Group | Dose Level B of Balovaptan | Placebo
Number analyzed (Participants) | 52 | 52
ms
  Day 14 0.75 hours Pre-dose | -0.1 [-1.89 to 1.64] | -0.6 [-2.35 to 1.18]
  Day 14 0.5 hours Pre-dose | -0.1 [-1.92 to 1.67] | 0.1 [-1.68 to 1.92]
  Day 14 0.25 hours Pre-dose: number analyzed (Participants) | 51 | 52
  Day 14 0.25 hours Pre-dose | 0.2 [-1.64 to 2.01] | -0.1 [-1.91 to 1.74]
  Day 14 0.5 hours Post-dose | -3.3 [-5.15 to -1.52] | -3.9 [-5.73 to -2.09]
  Day 14 1 hours Post-dose | -2.5 [-4.27 to -0.67] | -2.3 [-4.13 to -0.53]
  Day 14 2.5 hours Post-dose | -1.9 [-3.71 to -0.10] | -3.5 [-5.33 to -1.71]
  Day 14 4 hours Post-dose | -1.0 [-2.96 to 0.98] | -2.1 [-4.08 to -0.12]
  Day 14 8 hours Post-dose: number analyzed (Participants) | 51 | 52
  Day 14 8 hours Post-dose | -9.8 [-11.90 to -7.65] | -9.6 [-11.73 to -7.48]
  Day 14 12 hours Post-dose | -6.6 [-9.11 to -4.05] | -7.5 [-10.05 to -4.99]
  Day 14 24 hours Post-dose | -2.4 [-4.19 to -0.57] | -2.9 [-4.67 to -1.04]
Statistical Analysis 1: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QTcF (ms) at Day 14 0.75 Hours Pre-dose; LS Mean = 0.5, 90% CI 2-sided [-1.99 to 2.90], Standard Error of Mean 1.47
Statistical Analysis 2: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QTcF (ms) at Day 14 0.5 Hours Pre-dose; LS Mean = -0.2, 90% CI 2-sided [-2.73 to 2.24], Standard Error of Mean 1.50
Statistical Analysis 3: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QTcF (ms) at Day 14 0.25 Hours Pre-dose; LS Mean = 0.3, 90% CI 2-sided [-2.25 to 2.79], Standard Error of Mean 1.52
Statistical Analysis 4: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QTcF (ms) at Day 14 0.5 Hours Post-dose; LS Mean = 0.6, 90% CI 2-sided [-1.94 to 3.09], Standard Error of Mean 1.52
Statistical Analysis 5: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QTcF (ms) at Day 14 1 Hours Post-dose; LS Mean = -0.1, 90% CI 2-sided [-2.62 to 2.35], Standard Error of Mean 1.50
Statistical Analysis 6: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QTcF (ms) at Day 14 2.5 Hours Post-dose; LS Mean = 1.6, 90% CI 2-sided [-0.88 to 4.11], Standard Error of Mean 1.51
Statistical Analysis 7: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QTcF (ms) at Day 14 4 Hours Post-dose; LS Mean = 1.1, 90% CI 2-sided [-1.63 to 3.85], Standard Error of Mean 1.66
Statistical Analysis 8: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QTcF (ms) at Day 14 8 Hours Post-dose; LS Mean = -0.2, 90% CI 2-sided [-3.13 to 2.79], Standard Error of Mean 1.79
Statistical Analysis 9: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QTcF (ms) at Day 14 12 Hours Post-dose; LS Mean = 0.9, 90% CI 2-sided [-2.60 to 4.47], Standard Error of Mean 2.13
Statistical Analysis 10: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QTcF (ms) at Day 14 24 Hours Post-dose; LS Mean = 0.5, 90% CI 2-sided [-2.03 to 2.98], Standard Error of Mean 1.52

2. Secondary Outcome: Change-From-Baseline QTcF at Dose Level B Measured on 12-Lead ECGs Extracted From Continuous Recordings
Description: Change-from-baseline QTcF (ΔΔQTcF) at dose level B of balovaptan measured on 12-lead ECGs extracted from continuous recordings at the specified time points on Day 1.
Time Frame: Baseline (Predose Day 1), Day 1. (Each treatment period is 15 days.)
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: ms
Groups:
- Dose Level B of Balovaptan: Participants received dose level B of balovaptan.
Arm/Group | Dose Level B of Balovaptan | Placebo
Number analyzed (Participants) | 52 | 52
ms
  Day 1 0.5 hours Post-dose | -2.3 [-3.36 to -1.22] | -3.5 [-4.59 to -2.44]
  Day 1 1 hours Post-dose: number analyzed (Participants) | 52 | 51
  Day 1 1 hours Post-dose | -1.8 [-2.78 to -0.89] | -2.9 [-3.89 to -1.99]
  Day 1 2.5 hours Post-dose | -0.2 [-1.39 to 1.04] | -2.2 [-3.43 to -0.99]
  Day 1 4 hours Post-dose | 1.1 [-0.32 to 2.52] | -1.4 [-2.88 to -0.02]
  Day 1 8 hours Post-dose | -8.4 [-10.20 to -6.69] | -11.0 [-12.72 to -9.20]
  Day 1 12 hours Post-dose: number analyzed (Participants) | 51 | 52
  Day 1 12 hours Post-dose | -5.5 [-7.70 to -3.32] | -6.9 [-9.12 to -4.75]
  Day 1 24 hours Post-dose | -1.3 [-2.61 to -0.04] | -3.0 [-4.26 to -1.67]
Statistical Analysis 1: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QTcF (ms) at Day 1 0.5 Hours Post-dose; LS Mean = 1.2, 90% CI 2-sided [-0.19 to 2.64], Standard Error of Mean 0.86
Statistical Analysis 2: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QTcF (ms) at Day 1 1 Hours Post-dose; LS Mean = 1.1, 90% CI 2-sided [-0.12 to 2.33], Standard Error of Mean 0.74
Statistical Analysis 3: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QTcF (ms) at Day 1 2.5 Hours Post-dose; LS Mean = 2.0, 90% CI 2-sided [0.40 to 3.67], Standard Error of Mean 0.99
Statistical Analysis 4: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QTcF (ms) at Day 1 4 Hours Post-dose; LS Mean = 2.5, 90% CI 2-sided [0.60 to 4.49], Standard Error of Mean 1.18
Statistical Analysis 5: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QTcF (ms) at Day 1 8 Hours Post-dose; LS Mean = 2.5, 90% CI 2-sided [0.09 to 4.94], Standard Error of Mean 1.46
Statistical Analysis 6: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QTcF (ms) at Day 1 12 Hours Post-dose; LS Mean = 1.4, 90% CI 2-sided [-1.62 to 4.47], Standard Error of Mean 1.84
Statistical Analysis 7: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QTcF (ms) at Day 1 24 Hours Post-dose; LS Mean = 1.6, 90% CI 2-sided [-0.10 to 3.39], Standard Error of Mean 1.05

3. Secondary Outcome: Change-From-Baseline QTcF of Balovaptan at Dose Level A Measurred on 12-Lead ECGs Extracted From Continuous Recordings
Description: Change-from-baseline QTcF (ΔΔQTcF) at dose level A of balovaptan measured on 12-lead ECGs extracted from continuous recordings at the specified time points on Days 1 and 14.
Time Frame: Baseline (Predose Day 1), Day 1 and Day 14. (Each treatment period is 15 days.)
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: ms
Groups:
- Dose Level A of Balovaptan: Participants received dose level A of balovaptan.
Arm/Group | Dose Level A of Balovaptan | Placebo
Number analyzed (Participants) | 55 | 52
ms
  Day 1 0.5 hours Post-dose | -2.7 [-3.75 to -1.68] | -3.5 [-4.59 to -2.44]
  Day 1 1 hours Post-dose: number analyzed (Participants) | 55 | 51
  Day 1 1 hours Post-dose | -1.6 [-2.51 to -0.68] | -2.9 [-3.89 to -1.99]
  Day 1 2.5 hours Post-dose | -0.6 [-1.74 to 0.62] | -2.2 [-3.43 to -0.99]
  Day 1 4 hours Post-dose | -0.2 [-1.55 to 1.22] | -1.4 [-2.88 to -0.02]
  Day 1 8 hours Post-dose: number analyzed (Participants) | 54 | 52
  Day 1 8 hours Post-dose | -8.7 [-10.40 to -6.97] | -11.0 [-12.72 to -9.20]
  Day 1 12 hours Post-dose: number analyzed (Participants) | 54 | 52
  Day 1 12 hours Post-dose | -6.2 [-8.37 to -4.12] | -6.9 [-9.12 to -4.75]
  Day 1 24 hours Post-dose: number analyzed (Participants) | 54 | 52
  Day 1 24 hours Post-dose | -2.6 [-3.85 to -1.33] | -3.0 [-4.26 to -1.67]
  Day 14 0.75 hours Pre-dose: number analyzed (Participants) | 54 | 52
  Day 14 0.75 hours Pre-dose | -1.1 [-2.84 to 0.62] | -0.6 [-2.35 to 1.18]
  Day 14 0.5 hours Pre-dose: number analyzed (Participants) | 54 | 52
  Day 14 0.5 hours Pre-dose | -0.6 [-2.37 to 1.14] | 0.1 [-1.68 to 1.92]
  Day 14 0.25 hours Pre-dose: number analyzed (Participants) | 54 | 52
  Day 14 0.25 hours Pre-dose | 0.2 [-1.63 to 1.94] | -0.1 [-1.91 to 1.74]
  Day 14 0.5 hours Post-dose: number analyzed (Participants) | 54 | 52
  Day 14 0.5 hours Post-dose | -3.4 [-5.22 to -1.66] | -3.9 [-5.73 to -2.09]
  Day 14 1 hours Post-dose: number analyzed (Participants) | 54 | 52
  Day 14 1 hours Post-dose | -2.3 [-4.01 to -0.49] | -2.3 [-4.13 to -0.53]
  Day 14 2.5 hours Post-dose: number analyzed (Participants) | 54 | 52
  Day 14 2.5 hours Post-dose | -1.7 [-3.48 to 0.05] | -3.5 [-5.33 to -1.71]
  Day 14 4 hours Post-dose: number analyzed (Participants) | 54 | 52
  Day 14 4 hours Post-dose | -1.5 [-3.43 to 0.43] | -2.1 [-4.08 to -0.12]
  Day 14 8 hours Post-dose: number analyzed (Participants) | 54 | 52
  Day 14 8 hours Post-dose | -9.1 [-11.13 to -6.99] | -9.6 [-11.73 to -7.48]
  Day 14 12 hours Post-dose: number analyzed (Participants) | 54 | 52
  Day 14 12 hours Post-dose | -6.9 [-9.34 to -4.41] | -7.5 [-10.05 to -4.99]
  Day 14 24 hours Post-dose: number analyzed (Participants) | 54 | 52
  Day 14 24 hours Post-dose | -2.7 [-4.51 to -0.96] | -2.9 [-4.67 to -1.04]
Statistical Analysis 1: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QTcF (ms) at Day 1 0.5 Hours Post-dose; LS Mean = 0.8, 90% CI 2-sided [-0.60 to 2.20], Standard Error of Mean 0.85
Statistical Analysis 2: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QTcF (ms) at Day 1 1 Hours Post-dose; LS Mean = 1.3, 90% CI 2-sided [0.13 to 2.55], Standard Error of Mean 0.73
Statistical Analysis 3: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QTcF (ms) at Day 1 2.5 Hours Post-dose; LS Mean = 1.7, 90% CI 2-sided [0.04 to 3.27], Standard Error of Mean 0.98
Statistical Analysis 4: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QTcF (ms) at Day 1 4 Hours Post-dose; LS Mean = 1.3, 90% CI 2-sided [-0.64 to 3.20], Standard Error of Mean 1.16
Statistical Analysis 5: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QTcF (ms) at Day 1 8 Hours Post-dose; LS Mean = 2.3, 90% CI 2-sided [-0.13 to 4.67], Standard Error of Mean 1.45
Statistical Analysis 6: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QTcF (ms) at Day 1 12 Hours Post-dose; LS Mean = 0.7, 90% CI 2-sided [-2.31 to 3.70], Standard Error of Mean 1.82
Statistical Analysis 7: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QTcF (ms) at Day 1 24 Hours Post-dose; LS Mean = 0.4, 90% CI 2-sided [-1.35 to 2.10], Standard Error of Mean 1.04
Statistical Analysis 8: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QTcF (ms) at Day 14 0.75 Hours Pre-dose; LS Mean = -0.5, 90% CI 2-sided [-2.94 to 1.89], Standard Error of Mean 1.46
Statistical Analysis 9: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QTcF (ms) at Day 14 0.5 Hours Pre-dose; LS Mean = -0.7, 90% CI 2-sided [-3.19 to 1.72], Standard Error of Mean 1.48
Statistical Analysis 10: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QTcF (ms) at Day 14 0.25 Hours Pre-dose; LS Mean = 0.2, 90% CI 2-sided [-2.26 to 2.74], Standard Error of Mean 1.51
Statistical Analysis 11: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QTcF (ms) at Day 14 0.5 Hours Post-dose; LS Mean = 0.5, 90% CI 2-sided [-2.02 to 2.96], Standard Error of Mean 1.51
Statistical Analysis 12: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Equivalence — Placebo-corrected change-from-baseline QTcF (ms) at Day 14 1 Hours Post-dose; LS Mean = 0.1, 90% CI 2-sided [-2.39 to 2.54], Standard Error of Mean 1.49
Statistical Analysis 13: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QTcF (ms) at Day 14 2.5 Hours Post-dose; LS Mean = 1.8, 90% CI 2-sided [-0.67 to 4.28], Standard Error of Mean 1.50
Statistical Analysis 14: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QTcF (ms) at Day 14 4 Hours Post-dose; LS Mean = 0.6, 90% CI 2-sided [-2.11 to 3.31], Standard Error of Mean 1.64
Statistical Analysis 15: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QTcF (ms) at Day 14 8 Hours Post-dose; LS Mean = 0.5, 90% CI 2-sided [-2.38 to 3.47], Standard Error of Mean 1.76
Statistical Analysis 16: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QTcF (ms) at Day 14 12 Hours Post-dose; LS Mean = 0.6, 90% CI 2-sided [-2.85 to 4.14], Standard Error of Mean 2.11
Statistical Analysis 17: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QTcF (ms) at Day 14 24 Hours Post-dose; LS Mean = 0.1, 90% CI 2-sided [-2.36 to 2.60], Standard Error of Mean 1.50

4. Secondary Outcome: Change-From-Baseline Heart Rate Measured on 12-Lead ECGs Extracted From Continuous Recordings
Description: Change-from-baseline heart rate at dose level A and dose level B of balovaptan measured on 12-Lead ECGs extracted from continuous recordings on Days 1 and 14.
Time Frame: Baseline (Predose Day 1), Day 1 and Day 14. (Each treatment period is 15 days.)
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: bpm
Arm/Group | Dose Level A of Balovaptan | Dose Level B of Balovaptan | Placebo
Number analyzed (Participants) | 55 | 52 | 52
bpm
  Day 1 0.5 hours Post-dose | 0.2 [-0.54 to 0.91] | 0.5 [-0.24 to 1.25] | 0.4 [-0.34 to 1.17]
  Day 1 1 hours Post-dose: number analyzed (Participants) | 55 | 52 | 51
  Day 1 1 hours Post-dose | 0.1 [-0.64 to 0.87] | 0.0 [-0.78 to 0.78] | 0.2 [-0.61 to 0.97]
  Day 1 2.5 hours Post-dose | -0.4 [-1.29 to 0.54] | -0.3 [-1.28 to 0.60] | 0.1 [-0.85 to 1.04]
  Day 1 4 hours Post-dose | -0.4 [-1.35 to 0.47] | 0.3 [-0.64 to 1.24] | 0.1 [-0.83 to 1.05]
  Day 1 8 hours Post-dose: number analyzed (Participants) | 54 | 52 | 52
  Day 1 8 hours Post-dose | 4.8 [3.52 to 6.00] | 4.7 [3.43 to 5.97] | 5.4 [4.17 to 6.72]
  Day 1 12 hours Post-dose: number analyzed (Participants) | 54 | 51 | 52
  Day 1 12 hours Post-dose | 7.4 [6.02 to 8.80] | 7.9 [6.45 to 9.31] | 8.1 [6.69 to 9.54]
  Day 1 24 hours Post-dose: number analyzed (Participants) | 54 | 52 | 52
  Day 1 24 hours Post-dose | 2.2 [1.24 to 3.24] | 0.5 [-0.49 to 1.55] | 2.8 [1.75 to 3.80]
  Day 14 0.75 hours Pre-dose: number analyzed (Participants) | 54 | 52 | 52
  Day 14 0.75 hours Pre-dose | -0.6 [-1.81 to 0.64] | 0.9 [-0.34 to 2.16] | 1.6 [0.35 to 2.86]
  Day 14 0.5 hours Pre-dose: number analyzed (Participants) | 54 | 52 | 52
  Day 14 0.5 hours Pre-dose | -0.1 [-1.36 to 1.09] | 0.3 [-0.91 to 1.59] | 1.6 [0.32 to 2.82]
  Day 14 0.25 hours Pre-dose: number analyzed (Participants) | 54 | 51 | 52
  Day 14 0.25 hours Pre-dose | 0.3 [-0.94 to 1.62] | 1.0 [-0.32 to 2.30] | 1.8 [0.46 to 3.07]
  Day 14 0.5 hours Post-dose: number analyzed (Participants) | 54 | 52 | 52
  Day 14 0.5 hours Post-dose | 0.4 [-0.74 to 1.60] | 1.4 [0.16 to 2.55] | 2.0 [0.85 to 3.25]
  Day 14 1 hours Post-dose: number analyzed (Participants) | 54 | 52 | 52
  Day 14 1 hours Post-dose | 0.4 [-0.84 to 1.57] | 1.1 [-0.14 to 2.32] | 2.0 [0.82 to 3.28]
  Day 14 2.5 hours Post-dose: number analyzed (Participants) | 54 | 52 | 52
  Day 14 2.5 hours Post-dose | 0.6 [-0.70 to 1.88] | 1.2 [-0.07 to 2.56] | 2.5 [1.22 to 3.85]
  Day 14 4 hours Post-dose: number analyzed (Participants) | 54 | 52 | 52
  Day 14 4 hours Post-dose | 1.5 [0.27 to 2.67] | 1.8 [0.59 to 3.05] | 2.9 [1.63 to 4.09]
  Day 14 8 hours Post-dose: number analyzed (Participants) | 54 | 51 | 52
  Day 14 8 hours Post-dose | 5.2 [3.79 to 6.70] | 5.6 [4.08 to 7.07] | 6.3 [4.79 to 7.77]
  Day 14 12 hours Post-dose: number analyzed (Participants) | 54 | 52 | 52
  Day 14 12 hours Post-dose | 8.7 [7.31 to 10.01] | 9.2 [7.83 to 10.59] | 9.8 [8.41 to 11.17]
  Day 14 24 hours Post-dose: number analyzed (Participants) | 54 | 52 | 52
  Day 14 24 hours Post-dose | 2.3 [0.93 to 3.60] | 1.6 [0.21 to 2.94] | 3.3 [1.90 to 4.63]
Statistical Analysis 1: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline HR (bpm) at Day 1 0.5 Hours Post-dose; LS Mean = -0.2, 90% CI 2-sided [-1.20 to 0.73], Standard Error of Mean 0.59
Statistical Analysis 2: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline HR (bpm) at Day 1 1 Hours Post-dose; LS Mean = -0.1, 90% CI 2-sided [-1.08 to 0.96], Standard Error of Mean 0.62
Statistical Analysis 3: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline HR (bpm) at Day 1 2.5 Hours Post-dose; LS Mean = -0.5, 90% CI 2-sided [-1.73 to 0.78], Standard Error of Mean 0.76
Statistical Analysis 4: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline HR (bpm) at Day 1 4 Hours Post-dose; LS Mean = -0.6, 90% CI 2-sided [-1.80 to 0.70], Standard Error of Mean 0.75
Statistical Analysis 5: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline HR (bpm) at Day 1 8 Hours Post-dose; LS Mean = -0.7, 90% CI 2-sided [-2.42 to 1.05], Standard Error of Mean 1.05
Statistical Analysis 6: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline HR (bpm) at Day 1 12 Hours Post-dose; LS Mean = -0.7, 90% CI 2-sided [-2.66 to 1.24], Standard Error of Mean 1.18
Statistical Analysis 7: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline HR (bpm) at Day 1 24 Hours Post-dose; LS Mean = -0.5, 90% CI 2-sided [-1.91 to 0.85], Standard Error of Mean 0.83
Statistical Analysis 8: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline HR (bpm) at Day 14 0.75 Hours Pre-dose; LS Mean = -2.2, 90% CI 2-sided [-3.90 to -0.48], Standard Error of Mean 1.03
Statistical Analysis 9: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline HR (bpm) at Day 14 0.5 Hours Pre-dose; LS Mean = -1.7, 90% CI 2-sided [-3.41 to 0.00], Standard Error of Mean 1.03
Statistical Analysis 10: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline HR (bpm) at Day 14 0.25 Hours Pre-dose; LS Mean = -1.4, 90% CI 2-sided [-3.21 to 0.36], Standard Error of Mean 1.08
Statistical Analysis 11: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline HR (bpm) at Day 14 0.5 Hours Pre-dose; LS Mean = -1.6, 90% CI 2-sided [-3.25 to 0.01], Standard Error of Mean 0.98
Statistical Analysis 12: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline HR (bpm) at Day 14 1 Hours Post-dose; LS Mean = -1.7, 90% CI 2-sided [-3.36 to -0.01], Standard Error of Mean 1.01
Statistical Analysis 13: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline HR (bpm) at Day 14 2.5 Hours Post-dose; LS Mean = -1.9, 90% CI 2-sided [-3.75 to -0.14], Standard Error of Mean 1.09
Statistical Analysis 14: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline HR (bpm) at Day 14 4 Hours Post-dose; LS Mean = -1.4, 90% CI 2-sided [-3.06 to 0.29], Standard Error of Mean 1.01
Statistical Analysis 15: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline HR (bpm) at Day 14 8 Hours Post-dose; LS Mean = -1.0, 90% CI 2-sided [-3.08 to 1.01], Standard Error of Mean 1.24
Statistical Analysis 16: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline HR (bpm) at Day 14 12 Hours Post-dose; LS Mean = -1.1, 90% CI 2-sided [-3.03 to 0.76], Standard Error of Mean 1.14
Statistical Analysis 17: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline HR (bpm) at Day 14 24 Hours Post-dose; LS Mean = -1.0, 90% CI 2-sided [-2.87 to 0.87], Standard Error of Mean 1.13
Statistical Analysis 18: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline HR (bpm) at Day 1 0.5 Hours Post-dose; LS Mean = 0.1, 90% CI 2-sided [-0.89 to 1.07], Standard Error of Mean 0.59
Statistical Analysis 19: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline HR (bpm) at Day 1 1 Hours Post-dose; LS Mean = -0.2, 90% CI 2-sided [-1.21 to 0.86], Standard Error of Mean 0.62
Statistical Analysis 20: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline HR (bpm) at Day 1 2.5 Hours Post-dose; LS Mean = -0.4, 90% CI 2-sided [-1.71 to 0.83], Standard Error of Mean 0.77
Statistical Analysis 21: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline HR (bpm) at Day 1 4 Hours Post-dose; LS Mean = 0.2, 90% CI 2-sided [-1.07 to 1.46], Standard Error of Mean 0.76
Statistical Analysis 22: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline HR (bpm) at Day 1 8 Hours Post-dose; LS Mean = -0.8, 90% CI 2-sided [-2.50 to 1.00], Standard Error of Mean 1.06
Statistical Analysis 23: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline HR (bpm) at Day 1 12 Hours Post-dose; LS Mean = -0.2, 90% CI 2-sided [-2.22 to 1.74], Standard Error of Mean 1.19
Statistical Analysis 24: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline HR (bpm) at Day 1 24 Hours Post-dose; LS Mean = -2.2, 90% CI 2-sided [-3.63 to -0.85], Standard Error of Mean 0.84
Statistical Analysis 25: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline HR (bpm) at Day 14 0.75 Hours Pre-dose; LS Mean = -0.7, 90% CI 2-sided [-2.42 to 1.03], Standard Error of Mean 1.04
Statistical Analysis 26: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline Day 14 HR (bpm) at 0.5 Hours Pre-dose; LS Mean = -1.2, 90% CI 2-sided [-2.96 to 0.49], Standard Error of Mean 1.04
Statistical Analysis 27: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline HR (bpm) at Day 14 0.25 Hours Pre-dose; LS Mean = -0.8, 90% CI 2-sided [-2.58 to 1.02], Standard Error of Mean 1.09
Statistical Analysis 28: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline HR (bpm) at Day 14 0.5 Hours Post-dose; LS Mean = -0.7, 90% CI 2-sided [-2.34 to 0.95], Standard Error of Mean 0.99
Statistical Analysis 29: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline HR (bpm) at Day 14 1 Hours Post-dose; LS Mean = -1.0, 90% CI 2-sided [-2.65 to 0.73], Standard Error of Mean 1.02
Statistical Analysis 30: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline HR (bpm) at Day 14 2.5 Hours Post-dose; LS Mean = -1.3, 90% CI 2-sided [-3.11 to 0.53], Standard Error of Mean 1.10
Statistical Analysis 31: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline HR (bpm) at Day 14 4 Hours Post-dose; LS Mean = -1.0, 90% CI 2-sided [-2.73 to 0.66], Standard Error of Mean 1.02
Statistical Analysis 32: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline HR (bpm) at Day 14 8 Hours Post-dose; LS Mean = -0.7, 90% CI 2-sided [-2.77 to 1.37], Standard Error of Mean 1.25
Statistical Analysis 33: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline HR (bpm) at Day 14 12 Hours Post-dose; LS Mean = -0.6, 90% CI 2-sided [-2.50 to 1.33], Standard Error of Mean 1.15
Statistical Analysis 34: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline HR (bpm) at Day 14 24 Hours Post-dose; LS Mean = -1.7, 90% CI 2-sided [-3.57 to 0.20], Standard Error of Mean 1.14

5. Secondary Outcome: Change-From-Baseline PR Interval Measured on 12-Lead ECGs Extracted From Continuous Recordings
Description: Change-from-baseline PR interval at dose level A and dose level B of balovaptan measured on 12-Lead ECGs extracted from continuous recordings on Day 1 and 14.
Time Frame: Baseline (Predose Day 1), Day 1 and Day 14. (Each treatment period is 15 days.)
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: ms
Arm/Group | Dose Level A of Balovaptan | Dose Level B of Balovaptan | Placebo
Number analyzed (Participants) | 55 | 52 | 52
ms
  Day 1 0.5 hours Post-dose | -1.4 [-2.43 to -0.43] | -0.9 [-1.88 to 0.18] | -0.2 [-1.28 to 0.80]
  Day 1 1 hours Post-dose: number analyzed (Participants) | 55 | 52 | 51
  Day 1 1 hours Post-dose | -0.3 [-1.45 to 0.84] | -0.4 [-1.55 to 0.80] | -0.3 [-1.46 to 0.92]
  Day 1 2.5 hours Post-dose: number analyzed (Participants) | 55 | 51 | 52
  Day 1 2.5 hours Post-dose | -1.6 [-2.79 to -0.40] | -2.0 [-3.22 to -0.74] | -2.0 [-3.26 to -0.79]
  Day 1 4 hours Post-dose | -1.5 [-2.76 to -0.33] | -1.9 [-3.12 to -0.62] | -1.2 [-2.44 to 0.07]
  Day 1 8 hours Post-dose | -6.3 [-7.80 to -4.72] | -6.5 [-8.08 to -4.91] | -7.4 [-9.02 to -5.84]
  Day 1 12 hours Post-dose: number analyzed (Participants) | 55 | 50 | 52
  Day 1 12 hours Post-dose | -3.9 [-5.75 to -2.09] | -5.5 [-7.39 to -3.60] | -4.2 [-6.10 to -2.32]
  Day 1 24 hours Post-dose: number analyzed (Participants) | 54 | 52 | 52
  Day 1 24 hours Post-dose | -1.4 [-2.76 to -0.01] | -0.3 [-1.73 to 1.07] | -0.3 [-1.70 to 1.11]
  Day 14 0.75 hours Pre-dose: number analyzed (Participants) | 54 | 52 | 52
  Day 14 0.75 hours Pre-dose | 3.8 [1.84 to 5.69] | 4.5 [2.56 to 6.49] | 3.1 [1.17 to 5.10]
  Day 14 0.5 hours Pre-dose: number analyzed (Participants) | 54 | 52 | 52
  Day 14 0.5 hours Pre-dose | 4.1 [2.11 to 6.08] | 5.0 [2.97 to 7.02] | 3.8 [1.75 to 5.81]
  Day 14 0.25 hours Pre-dose: number analyzed (Participants) | 54 | 51 | 52
  Day 14 0.25 hours Pre-dose | 3.2 [1.24 to 5.21] | 4.5 [2.46 to 6.52] | 3.0 [0.94 to 5.00]
  Day 14 0.5 hours Post-dose: number analyzed (Participants) | 54 | 52 | 52
  Day 14 0.5 hours Post-dose | 2.9 [0.67 to 5.11] | 2.7 [0.44 to 4.98] | 2.9 [0.64 to 5.18]
  Day 14 1 hours Post-dose: number analyzed (Participants) | 54 | 52 | 52
  Day 14 1 hours Post-dose | 3.1 [0.99 to 5.12] | 2.1 [-0.04 to 4.19] | 2.6 [0.49 to 4.72]
  Day 14 2.5 hours Post-dose: number analyzed (Participants) | 54 | 52 | 52
  Day 14 2.5 hours Post-dose | 0.2 [-1.85 to 2.23] | 1.8 [-0.25 to 3.92] | 0.7 [-1.36 to 2.82]
  Day 14 4 hours Post-dose: number analyzed (Participants) | 54 | 52 | 52
  Day 14 4 hours Post-dose | -0.9 [-2.95 to 1.05] | 0.9 [-1.10 to 2.99] | -0.2 [-2.29 to 1.81]
  Day 14 8 hours Post-dose: number analyzed (Participants) | 54 | 52 | 52
  Day 14 8 hours Post-dose | -5.1 [-6.90 to -3.22] | -3.7 [-5.55 to -1.79] | -4.3 [-6.23 to -2.46]
  Day 14 12 hours Post-dose: number analyzed (Participants) | 54 | 52 | 52
  Day 14 12 hours Post-dose | -2.8 [-4.65 to -0.89] | -0.9 [-2.86 to 0.99] | -4.2 [-6.14 to -2.29]
  Day 14 24 hours Post-dose: number analyzed (Participants) | 54 | 52 | 52
  Day 14 24 hours Post-dose | 0.9 [-0.99 to 2.84] | 3.1 [1.18 to 5.08] | 1.1 [-0.82 to 3.08]
Statistical Analysis 1: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline PR (ms) at Day 1 0.5 Hours Post-dose; LS Mean = -1.2, 90% CI 2-sided [-2.56 to 0.17], Standard Error of Mean 0.83
Statistical Analysis 2: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline PR (ms) at Day 1 1 Hours Post-dose; LS Mean = 0.0, 90% CI 2-sided [-1.62 to 1.55], Standard Error of Mean 0.96
Statistical Analysis 3: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline PR (ms) at Day 1 2.5 Hours Post-dose; LS Mean = 0.4, 90% CI 2-sided [-1.22 to 2.09], Standard Error of Mean 1.00
Statistical Analysis 4: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline PR (ms) at Day 1 4 Hours Post-dose; LS Mean = -0.4, 90% CI 2-sided [-2.04 to 1.33], Standard Error of Mean 1.02
Statistical Analysis 5: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline PR (ms) at Day 1 8 Hours Post-dose; LS Mean = 1.2, 90% CI 2-sided [-1.00 to 3.33], Standard Error of Mean 1.31
Statistical Analysis 6: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline PR (ms) at Day 1 12 Hours Post-dose; LS Mean = 0.3, 90% CI 2-sided [-2.30 to 2.88], Standard Error of Mean 1.56
Statistical Analysis 7: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline PR (ms) at Day 1 24 Hours Post-dose; LS Mean = -1.1, 90% CI 2-sided [-3.00 to 0.81], Standard Error of Mean 1.15
Statistical Analysis 8: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline PR (ms) at Day 14 0.75 Hours Pre-dose; LS Mean = 0.6, 90% CI 2-sided [-2.08 to 3.35], Standard Error of Mean 1.64
Statistical Analysis 9: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline PR (ms) at Day 14 0.5 Hours Pre-dose; LS Mean = 0.3, 90% CI 2-sided [-2.48 to 3.12], Standard Error of Mean 1.69
Statistical Analysis 10: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline PR (ms) at Day 14 0.25 Hours Pre-dose; LS Mean = 0.3, 90% CI 2-sided [-2.55 to 3.06], Standard Error of Mean 1.69
Statistical Analysis 11: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline PR (ms) at Day 14 0.5 Hours Post-dose; LS Mean = 0.0, 90% CI 2-sided [-3.17 to 3.12], Standard Error of Mean 1.90
Statistical Analysis 12: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline PR (ms) at Day 14 1 Hours Post-dose; LS Mean = 0.5, 90% CI 2-sided [-2.47 to 3.37], Standard Error of Mean 1.77
Statistical Analysis 13: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline PR (ms) at Day 14 2.5 Hours Post-dose; LS Mean = -0.5, 90% CI 2-sided [-3.42 to 2.34], Standard Error of Mean 1.74
Statistical Analysis 14: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline PR (ms) at Day 14 4 Hours Post-dose; LS Mean = -0.7, 90% CI 2-sided [-3.54 to 2.12], Standard Error of Mean 1.71
Statistical Analysis 15: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline PR (ms) at Day 14 8 Hours Post-dose; LS Mean = -0.7, 90% CI 2-sided [-3.31 to 1.88], Standard Error of Mean 1.57
Statistical Analysis 16: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline PR (ms) at Day 14 12 Hours Post-dose; LS Mean = 1.4, 90% CI 2-sided [-1.21 to 4.09], Standard Error of Mean 1.60
Statistical Analysis 17: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline PR (ms) at Day 14 24 Hours Post-dose; LS Mean = -0.2, 90% CI 2-sided [-2.90 to 2.49], Standard Error of Mean 1.63
Statistical Analysis 18: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline PR (ms) at Day 1 0.5 Hours Post-dose; LS Mean = -0.6, 90% CI 2-sided [-2.00 to 0.77], Standard Error of Mean 0.84
Statistical Analysis 19: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline PR (ms) at Day 1 1 Hours Post-dose; LS Mean = -0.1, 90% CI 2-sided [-1.71 to 1.50], Standard Error of Mean 0.97
Statistical Analysis 20: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline PR (ms) at Day 1 2.5 Hours Post-dose; LS Mean = 0.0, 90% CI [-1.64 to 1.73], Standard Error of Mean 1.02
Statistical Analysis 21: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline PR (ms) at Day 1 4 Hours Post-dose; LS Mean = -0.7, 90% CI 2-sided [-2.39 to 1.02], Standard Error of Mean 1.03
Statistical Analysis 22: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline PR (ms) at Day 1 8 Hours Post-dose; LS Mean = 0.9, 90% CI 2-sided [-1.26 to 3.13], Standard Error of Mean 1.33
Statistical Analysis 23: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline PR (ms) at Day 1 12 Hours Post-dose; LS Mean = -1.3, 90% CI [-3.92 to 1.35], Standard Error of Mean 1.59
Statistical Analysis 24: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline PR (ms) at Day 1 24 Hours Post-dose; LS Mean = 0.0, 90% CI 2-sided [-1.96 to 1.89], Standard Error of Mean 1.16
Statistical Analysis 25: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline PR (ms) at Day 14 0.75 Hours Pre-dose; LS Mean = 1.4, 90% CI 2-sided [-1.34 to 4.13], Standard Error of Mean 1.65
Statistical Analysis 26: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline PR (ms) at Day 14 0.5 Hours Pre-dose; LS Mean = 1.2, 90% CI 2-sided [-1.61 to 4.05], Standard Error of Mean 1.71
Statistical Analysis 27: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline PR (ms) at Day 14 0.25 Hours Pre-dose; LS Mean = 1.5, 90% CI 2-sided [-1.32 to 4.35], Standard Error of Mean 1.71
Statistical Analysis 28: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline PR (ms) at Day 14 0.5 Hours Post-dose; LS Mean = -0.2, 90% CI 2-sided [-3.38 to 2.97], Standard Error of Mean 1.92
Statistical Analysis 29: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline PR (ms) at Day 14 1 Hours Pre-dose; LS Mean = -0.5, 90% CI [-3.48 to 2.42], Standard Error of Mean 1.78
Statistical Analysis 30: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline PR (ms) at Day 14 2.5 Hours Post-dose; LS Mean = 1.1, 90% CI 2-sided [-1.81 to 4.02], Standard Error of Mean 1.76
Statistical Analysis 31: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline PR (ms) at Day 14 4 Hours Post-dose; LS Mean = 1.2, 90% CI 2-sided [-1.67 to 4.04], Standard Error of Mean 1.72
Statistical Analysis 32: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline PR (ms) at Day 14 8 Hours Post-dose; LS Mean = 0.7, 90% CI 2-sided [-1.95 to 3.29], Standard Error of Mean 1.58
Statistical Analysis 33: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline PR (ms) at Day 14 12 Hours Post-dose; LS Mean = 3.3, 90% CI 2-sided [0.60 to 5.96], Standard Error of Mean 1.62
Statistical Analysis 34: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline PR (ms) at Day 14 24 Hours Post-dose; LS Mean = 2.0, 90% CI 2-sided [-0.72 to 4.72], Standard Error of Mean 1.64

6. Secondary Outcome: Change-From-Baseline QRS Interval Measured on 12-Lead ECGs Extracted From Continuous Recordings
Description: Change-from-baseline QRS interval at dose level A and dose level B of balovapton measured on 12-Lead ECGs extracted from continuous recordings on Days 1 and 14.
Time Frame: Baseline (Predose Day 1), Day 1 and Day 14. (Each treatment period is 15 days.)
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: ms
Arm/Group | Dose Level A of Balovaptan | Dose Level B of Balovaptan | Placebo
Number analyzed (Participants) | 55 | 52 | 52
ms
  Day 1 0.5 hours Post-dose | -0.1 [-0.25 to 0.01] | -0.1 [-0.22 to 0.05] | 0.0 [-0.15 to 0.12]
  Day 1 1 hours Post-dose: number analyzed (Participants) | 55 | 52 | 51
  Day 1 1 hours Post-dose | 0.1 [-0.06 to 0.20] | 0.1 [-0.05 to 0.22] | -0.1 [-0.22 to 0.05]
  Day 1 2.5 hours Post-dose: number analyzed (Participants) | 55 | 51 | 52
  Day 1 2.5 hours Post-dose | 0.00 [-0.13 to 0.17] | 0.00 [-0.17 to 0.14] | 0.1 [-0.05 to 0.26]
  Day 1 4 hours Post-dose | 0.0 [-0.17 to 0.14] | 0.1 [-0.02 to 0.31] | 0.0 [-0.14 to 0.19]
  Day 1 8 hours Post-dose | -0.5 [-0.83 to -0.16] | -0.3 [-0.66 to 0.03] | -0.4 [-0.74 to -0.05]
  Day 1 12 hours Post-dose: number analyzed (Participants) | 55 | 50 | 52
  Day 1 12 hours Post-dose | -0.2 [-0.58 to 0.26] | 0.2 [-0.25 to 0.63] | -0.1 [-0.55 to 0.32]
  Day 1 24 hours Post-dose: number analyzed (Participants) | 54 | 52 | 52
  Day 1 24 hours Post-dose | 0.0 [-0.22 to 0.15] | 0.1 [-0.04 to 0.33] | -0.2 [-0.37 to 0.01]
  Day 14 0.75 hours Pre-dose: number analyzed (Participants) | 54 | 52 | 52
  Day 14 0.75 hours Pre-dose | 0.4 [0.03 to 0.79] | 0.6 [0.18 to 0.95] | 0.2 [-0.18 to 0.60]
  Day 14 0.5 hours Pre-dose: number analyzed (Participants) | 54 | 52 | 52
  Day 14 0.5 hours Pre-dose | 0.4 [0.03 to 0.79] | 0.5 [0.08 to 0.86] | 0.0 [-0.35 to 0.42]
  Day 14 0.25 hours Pre-dose: number analyzed (Participants) | 54 | 51 | 52
  Day 14 0.25 hours Pre-dose | 0.5 [0.15 to 0.92] | 0.5 [0.12 to 0.91] | 0.00 [-0.37 to 0.42]
  Day 14 0.5 hours Post-dose: number analyzed (Participants) | 54 | 52 | 52
  Day 14 0.5 hours Post-dose | 0.5 [0.10 to 0.87] | 0.5 [0.09 to 0.86] | 0.2 [-0.19 to 0.59]
  Day 14 1 hours Post-dose: number analyzed (Participants) | 54 | 52 | 52
  Day 14 1 hours Post-dose | 0.6 [0.18 to 0.94] | 0.6 [0.21 to 0.98] | 0.2 [-0.19 to 0.58]
  Day 14 2.5 hours Post-dose: number analyzed (Participants) | 54 | 52 | 52
  Day 14 2.5 hours Post-dose | 0.5 [0.12 to 0.89] | 0.4 [-0.04 to 0.75] | 0.0 [-0.35 to 0.43]
  Day 14 4 hours Post-dose: number analyzed (Participants) | 54 | 52 | 52
  Day 14 4 hours Post-dose | 0.4 [0.00 to 0.79] | 0.7 [0.25 to 1.06] | 0.0 [-0.39 to 0.42]
  Day 14 8 hours Post-dose: number analyzed (Participants) | 54 | 52 | 52
  Day 14 8 hours Post-dose | 0.1 [-0.38 to 0.62] | 0.4 [-0.14 to 0.88] | -0.3 [-0.77 to 0.25]
  Day 14 12 hours Post-dose: number analyzed (Participants) | 54 | 52 | 52
  Day 14 12 hours Post-dose | 0.6 [0.06 to 1.15] | 0.6 [0.06 to 1.17] | 0.3 [-0.23 to 0.89]
  Day 14 24 hours Post-dose: number analyzed (Participants) | 54 | 52 | 52
  Day 14 24 hours Post-dose | 0.6 [0.15 to 0.98] | 0.5 [0.07 to 0.91] | 0.00 [-0.38 to 0.46]
Statistical Analysis 1: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QRS (ms) at Day 1 0.5 Hours Post-dose; LS Mean = -0.1, 90% CI 2-sided [-0.29 to 0.07], Standard Error of Mean 0.11
Statistical Analysis 2: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QRS (ms) at Day 1 1 Hours Post-dose; LS Mean = 0.2, 90% CI 2-sided [-0.02 to 0.34], Standard Error of Mean 0.11
Statistical Analysis 3: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline (ms) at QRS Day 1 2.5 Hours Post-dose; LS Mean = -0.1, 90% CI 2-sided [-0.30 to 0.12], Standard Error of Mean 0.13
Statistical Analysis 4: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QRS (ms) at Day 1 4 Hours Post-dose; LS Mean = 0.0, 90% CI 2-sided [-0.26 to 0.18], Standard Error of Mean 0.13
Statistical Analysis 5: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QRS (ms) at Day 1 8 Hours Post-dose; LS Mean = -0.1, 90% CI 2-sided [-0.57 to 0.38], Standard Error of Mean 0.29
Statistical Analysis 6: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QRS (ms) at Day 1 12 Hours Post-dose; LS Mean = 0.0, 90% CI 2-sided [-0.65 to 0.56], Standard Error of Mean 0.37
Statistical Analysis 7: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QRS (ms) at Day 1 24 Hours Post-dose; LS Mean = 0.1, 90% CI [-0.11 to 0.40], Standard Error of Mean 0.15
Statistical Analysis 8: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QRS (ms) at Day 14 0.75 Hours Pre-dose; LS Mean = 0.2, 90% CI 2-sided [-0.34 to 0.74], Standard Error of Mean 0.33
Statistical Analysis 9: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QRS (ms) at Day 14 0.5 Hours Pre-dose; LS Mean = 0.4, 90% CI 2-sided [-0.17 to 0.91], Standard Error of Mean 0.33
Statistical Analysis 10: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QRS (ms) at Day 14 0.25 Hours Pre-dose; LS Mean = 0.5, 90% CI 2-sided [-0.04 to 1.05], Standard Error of Mean 0.33
Statistical Analysis 11: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QRS (ms) at Day 14 0.5 Hours Post-dose; LS Mean = 0.3, 90% CI 2-sided [-0.26 to 0.82], Standard Error of Mean 0.33
Statistical Analysis 12: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QRS (ms) at Day 14 1 Hours Post-dose; LS Mean = 0.4, 90% CI 2-sided [-0.18 to 0.90], Standard Error of Mean 032
Statistical Analysis 13: Comparison: Dose Level A of Balovaptan vs Placebo; Placebo-corrected change-from-baseline QRS (ms) at Day 14 2.5 Hours Post-dose; Test type: Other; LS Mean = 0.5, 90% CI 2-sided [-0.08 to 1.00], Standard Error of Mean 0.33
Statistical Analysis 14: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QRS (ms) at Day 14 4 Hours Post-dose; LS Mean = 0.4, 90% CI 2-sided [-0.19 to 0.94], Standard Error of Mean 0.34
Statistical Analysis 15: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QRS (ms) at Day 14 8 Hours Post-dose; LS Mean = 0.4, 90% CI 2-sided [-0.33 to 1.10], Standard Error of Mean 0.43
Statistical Analysis 16: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QRS (ms) at Day 14 12 Hours Post-dose; LS Mean = 0.3, 90% CI 2-sided [-0.50 to 1.06], Standard Error of Mean 0.47
Statistical Analysis 17: Comparison: Dose Level A of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QRS (ms) at Day 14 24 Hours Post-dose; LS Mean = 0.5, 90% CI 2-sided [-0.06 to 1.11], Standard Error of Mean 0.35
Statistical Analysis 18: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QRS (ms) at Day 1 0.5 Hours Post-dose; LS Mean = -0.1, 90% CI 2-sided [-0.25 to 0.11], Standard Error of Mean 0.11
Statistical Analysis 19: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QRS (ms) at Day 1 1 Hours Post-dose; LS Mean = 0.2, 90% CI 2-sided [0.00 to 0.36], Standard Error of Mean 0.11
Statistical Analysis 20: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QRS (ms) at Day 1 2.5 Hours Post-dose; LS Mean = -0.1, 90% CI 2-sided [-0.34 to 0.09], Standard Error of Mean 0.13
Statistical Analysis 21: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QRS (ms) at Day 1 4 Hours Post-dose; LS Mean = 0.1, 90% CI 2-sided [-0.10 to 0.34], Standard Error of Mean 0.13
Statistical Analysis 22: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QRS (ms) at Day 1 8 Hours Post-dose; LS Mean = 0.1, 90% CI 2-sided [-0.40 to 0.57], Standard Error of Mean 0.29
Statistical Analysis 23: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QRS (ms) at Day 1 12 Hours Post-dose; LS Mean = 0.3, 90% CI 2-sided [-0.31 to 0.93], Standard Error of Mean 0.37
Statistical Analysis 24: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QRS (ms) at Day 1 24 Hours Post-dose; LS Mean = 0.3, 90% CI 2-sided [0.07 to 0.58], Standard Error of Mean 0.16
Statistical Analysis 25: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QRS (ms) at Day 14 0.75 Hours Pre-dose; LS Mean = 0.4, 90% CI 2-sided [-0.19 to 0.90], Standard Error of Mean 0.33
Statistical Analysis 26: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QRS (ms) at Day 14 0.5 Hours Pre-dose; LS Mean = 0.4, 90% CI 2-sided [-0.11 to 0.98], Standard Error of Mean 0.33
Statistical Analysis 27: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QRS (ms) at Day 14 0.25 Hours Pre-dose; LS Mean = 0.5, 90% CI 2-sided [-0.06 to 1.05], Standard Error of Mean 0.33
Statistical Analysis 28: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QRS (ms) at Day 14 0.5 Hours Post-dose; LS Mean = 0.3, 90% CI 2-sided [-0.27 to 0.82], Standard Error of Mean 0.33
Statistical Analysis 29: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QRS (ms) at Day 14 1 Hours Post-dose; LS Mean = 0.4, 90% CI 2-sided [-0.14 to 0.94], Standard Error of Mean 0.33
Statistical Analysis 30: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QRS (ms) at Day 14 2.5 Hours Post-dose; LS Mean = 0.3, 90% CI 2-sided [-0.24 to 0.86], Standard Error of Mean 0.33
Statistical Analysis 31: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QRS (ms) at Day 14 4 Hours Post-dose; LS Mean = 0.6, 90% CI 2-sided [0.07 to 1.20], Standard Error of Mean 0.34
Statistical Analysis 32: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QRS (ms) at Day 14 8 Hours Post-dose; LS Mean = 0.6, 90% CI 2-sided [-0.10 to 1.35], Standard Error of Mean 0.44
Statistical Analysis 33: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QRS (ms) at Day 14 12 Hours Post-dose; LS Mean = 0.3, 90% CI 2-sided [-0.50 to 1.07], Standard Error of Mean 0.48
Statistical Analysis 34: Comparison: Dose Level B of Balovaptan vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QRS (ms) at Day 14 24 Hours Post-dose; LS Mean = 0.5, 90% CI 2-sided [-0.14 to 1.04], Standard Error of Mean 0.36

7. Secondary Outcome: Number of Categorical Outliers for QTcF
Description: The number (percentage) of categorical outliers were participants who had increases in absolute QTcF values > 450 and ≤ 480 ms, > 480 and ≤ 500 ms, or > 500 ms.
Time Frame: Up to approximately 20 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level A of Balovaptan | Dose Level B of Balovaptan | Placebo
Number analyzed (Participants) | 55 | 52 | 52
Participants
  QTcF>450 and <=480 ms | 0 | 1 | 0
  QTcF>480 and <=500 ms | 0 | 0 | 00
  QTcF>500 ms | 0 | 0 | 0

8. Secondary Outcome: Number of Categorical Outliers for HR
Description: Number (percentage) of categorical outliers were participants with a decrease in HR from pre-dose baseline > 25% to a HR < 50 bpm; and increase in HR from pre-dose baseline > 25% to a HR > 100 bpm.
Time Frame: Up to approximately 20 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Dose Level A of Balovaptan | Dose Level B of Balovaptan
Number analyzed (Participants) | 52 | 55 | 52
Participants
  HR < 50 (bpm) with a decrease in ΔHR > 25% | 0 | 0 | 0
  HR > 100 (bpm) with an increase in ΔHR > 25% | 0 | 0 | 0

9. Secondary Outcome: Number of Categorical Outliers for PR
Description: PR outliers criteria is as an increase of PR from baseline >25% resulting in PR >200 ms.
Time Frame: Up to approximately 20 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level A of Balovaptan | Dose Level B of Balovaptan | Placebo
Number analyzed (Participants) | 55 | 52 | 52
Participants | 0 | 0 | 0

10. Secondary Outcome: Number of Categorical Outliers for QRS
Description: QRS outlier criteria is an increase of QRS from baseline >25% resulting in QRS >120 ms.
Time Frame: Up to approximately 20 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Dose Level A of Balovaptan: All participants received Treatment A and Treatment B and either Treatment C or Treatment D.
Arm/Group | Dose Level A of Balovaptan | Dose Level B of Balovaptan | Placebo
Number analyzed (Participants) | 55 | 52 | 52
Participants | 0 | 0 | 0

11. Secondary Outcome: Number of Treatment Emergent Changes of T-Wave Morphology
Description: Number (%) of participants falling into each of the T-wave categories: Normal (+), Flat, Notched (+), Biphasic, Normal (-), Notched (-).
Time Frame: Up to approximately 20 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level A of Balovaptan | Dose Level B of Balovaptan | Placebo
Number analyzed (Participants) | 55 | 52 | 52
Participants
  Flat T-wave | 0 | 1 | 1
  Notched T-wave (+) | 0 | 0 | 0
  Biphasic T-wave | 0 | 1 | 0
  Normal T-wave (-) | 0 | 0 | 0
  Notched T-wave (-) | 0 | 0 | 0

12. Secondary Outcome: Number of Treatment Emergent Changes of U-Wave Presence
Description: Number (percentage) of participants with treatment emergent changes of U-wave presence.
Time Frame: Up to approximately 20 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level A of Balovaptan | Dose Level B of Balovaptan | Placebo
Number analyzed (Participants) | 55 | 52 | 52
Participants | 0 | 0 | 0

13. Secondary Outcome: Tmax of Balovaptan
Time Frame: Day 1 and Day 14. (Each treatment period is 15 days.)
Population: PK population included all participants who received at least 1 dose of investigational product and had at least 1 evaluable pharmacokinetic (PK) plasma concentration for any of balovaptan, M2 and M3 (and moxifloxacin, when applicable).
Measure: Median (Full Range); unit: h
Arm/Group | Dose Level A of Balovaptan | Dose Level B of Balovaptan
Number analyzed (Participants) | 55 | 52
h
  Day 1 | 2.50 [1.00 to 8.00] | 1.00 [0.50 to 4.00]
  Day 14: number analyzed (Participants) | 54 | 52
  Day 14 | 1.00 [1.00 to 8.00] | 1.00 [0.50 to 2.50]

14. Secondary Outcome: Tmax of M2 Metabolite
Time Frame: Day 1 and Day 14. (Each treatment period is 15 days.)
Population: as for outcome 13
Measure: Median (Full Range); unit: h
Arm/Group | Dose Level A of Balovaptan | Dose Level B of Balovaptan
Number analyzed (Participants) | 55 | 52
h
  Day 1 | 23.92 [12.00 to 23.95] | 23.92 [12.00 to 23.95]
  Day 14: number analyzed (Participants) | 54 | 52
  Day 14 | 6.00 [0.50 to 23.83] | 6.00 [0.50 to 12.00]

15. Secondary Outcome: Tmax M3 Metabolite
Time Frame: Day 1 and Day 14. (Each treatment period is 15 days.)
Population: as for outcome 13
Measure: Median (Full Range); unit: h
Arm/Group | Dose Level A of Balovaptan | Dose Level B of Balovaptan
Number analyzed (Participants) | 55 | 52
h
  Day 1 | 23.92 [6.00 to 23.95] | 8.00 [1.00 to 23.95]
  Day 14: number analyzed (Participants) | 54 | 52
  Day 14 | 4.00 [0.50 to 8.00] | 4.01 [0.50 to 8.10]

16. Secondary Outcome: Cmax of Balovaptan
Time Frame: Day 1 and Day 14. (Each treatment period is 15 days.)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dose Level A of Balovaptan | Dose Level B of Balovaptan
Number analyzed (Participants) | 55 | 52
ng/mL
  Day 1 | 32.5 (11.84) | 362.7 (122.47)
  Day 14: number analyzed (Participants) | 54 | 52
  Day 14 | 89.8 (28.98) | 613.4 (191.95)

17. Secondary Outcome: Cmax of M2 Metabolite
Time Frame: Day 1 and Day 14. (Each treatment period is 15 days.)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dose Level A of Balovaptan | Dose Level B of Balovaptan
Number analyzed (Participants) | 55 | 52
ng/mL
  Day 1 | 5.69 (1.828) | 42.75 (11.965)
  Day 14: number analyzed (Participants) | 54 | 52
  Day 14 | 24.77 (6.057) | 152.83 (40.855)

18. Secondary Outcome: Cmax of M3 Metabolite
Time Frame: Day 1 and Day 14. (Each treatment period is 15 days.)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dose Level A of Balovaptan | Dose Level B of Balovaptan
Number analyzed (Participants) | 55 | 52
ng/mL
  Day 1 | 6.83 (1.697) | 71.12 (17.615)
  Day 14: number analyzed (Participants) | 54 | 52
  Day 14 | 1005.2 (233.87) | 5456.9 (1253.40)

19. Secondary Outcome: AUC0-24 of Balovaptan
Time Frame: Day 1 and Day 14 (Each treatment period is 15 days.)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Dose Level A of Balovaptan | Dose Level B of Balovaptan
Number analyzed (Participants) | 55 | 52
h*ng/mL
  Day 1 | 440.7 (121.92) | 3524.8 (956.14)
  Day 14: number analyzed (Participants) | 54 | 52
  Day 14 | 1127.6 (372.72) | 6377.9 (2149.62)

20. Secondary Outcome: AUC0-24 of M2 Metabolite
Time Frame: Day 1 and Day 14 (Each treatment period is 15 days.)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Dose Level A of Balovaptan | Dose Level B of Balovaptan
Number analyzed (Participants) | 54 | 52
h*ng/mL
  Day 1 | 90.8 (30.55) | 766.6 (222.20)
  Day 14 | 527.5 (123.23) | 3127.0 (807.15)

21. Secondary Outcome: AUC0-24 of M3 Metabolite
Time Frame: Day 1 and Day 14 (Each treatment period is 15 days.)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Dose Level A of Balovaptan | Dose Level B of Balovaptan
Number analyzed (Participants) | 55 | 52
h*ng/mL
  Day 1: number analyzed (Participants) | 54 | 52
  Day 1 | 131.2 (37.49) | 1404.2 (344.31)
  Day 14: number analyzed (Participants) | 54 | 52
  Day 14 | 1005.2 (233.87) | 5456.9 (1253.40)

22. Secondary Outcome: Tmax of Moxifloxacin
Time Frame: Days 2 (Treatment C) or 15 (Treatment D). (Each treatment period is 15 days.)
Population: as for outcome 13
Measure: Median (Full Range); unit: h
Groups:
- Treatment C: Participants in Treatment C received 400 mg of Moxifloxacin on Day 2.
- Treatment D: Participants in Treatment D received 400 mg of Moxifloxacin on Day 15.
Arm/Group | Treatment C | Treatment D
Number analyzed (Participants) | 26 | 26
h | 2.50 [0.50 to 4.02] | 1.78 [0.50 to 4.02]

23. Secondary Outcome: Cmax of Moxifloxacin
Time Frame: Days 2 (Treatment C) or 15 (Treatment D) (Each treatment period is 15 days.)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Treatment C | Treatment D
Number analyzed (Participants) | 26 | 26
ng/mL | 2056.9 (437.64) | 2058.8 (525.99)

24. Secondary Outcome: AUC0-24 of Moxifloxacin
Time Frame: Days 2 (Treatment C) or 15 (Treatment D) (Each treatment period is 15 days.)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Treatment C | Treatment D
Number analyzed (Participants) | 26 | 26
h*ng/mL | 22503.9 (4103.73) | 24103.1 (5169.94)

25. Secondary Outcome: Predicted ΔΔQTcF Interval at Geometric Mean Peak Concentrations at Tmax of Balovaptan From Concentration-QTc Analysis
Time Frame: Baseline, Day 14. (Each treatment period is 15 days.)
Population: PK/QTc population included all participants who were in both the QT/QTc and PK populations with at least 1 pair of post-dose PK and QTcF data from the same time point.
Measure: Geometric Mean (90% Confidence Interval); unit: ms
Groups:
- Dose A of Balovaptan: Participants received dose A of Balovaptan.
- Dose B of Balovaptan: Participants received dose B of balovaptan
Arm/Group | Dose A of Balovaptan | Dose B of Balovaptan
Number analyzed (Participants) | 55 | 52
ms | 1.06 [-0.20 to 2.31] | 0.70 [-1.49 to 2.88]

26. Secondary Outcome: Predicted ΔΔQTcF Interval at Geometric Mean Peak Concentrations at Tmax of M2 From Concentration-QTc Analysis
Time Frame: Baseline, Day 14. (Each treatment period is 15 days.)
Population: as for outcome 25
Measure: Geometric Mean (90% Confidence Interval); unit: ms
Arm/Group | Dose Level A of Balovaptan | Dose Level B of Balovaptan
Number analyzed (Participants) | 55 | 52
ms | 1.01 [-0.30 to 2.31] | 0.27 [-2.47 to 3.02]

27. Secondary Outcome: Predicted ΔΔQTcF Interval at Geometric Mean Peak Concentration for M3 From Concentration-QTc Analysis
Time Frame: Baseline, Day 14. (Each treatment period is 15 days.)
Population: as for outcome 25
Measure: Geometric Mean (90% Confidence Interval); unit: ms
Arm/Group | Dose Level A of Balovaptan | Dose Level B of Balovaptan
Number analyzed (Participants) | 55 | 52
ms | 1.05 [-0.17 to 2.27] | 0.23 [-2.38 to 2.83]

28. Secondary Outcome: Change-From-Baseline QTcF Measured on 12 Lead ECGs Extracted From Continuous Records
Time Frame: Baseline, Day 15. (Each treatment period is 15 days.)
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: ms
Groups:
- Moxifloxacin: Participants received 400 mg of moxifloxacin
Arm/Group | Moxifloxacin | Placebo
Number analyzed (Participants) | 52 | 52
ms
  0.5 hours Post-dose | -2.0 [-4.01 to 0.02] | -3.2 [-5.21 to -1.18]
  1 hours Post-dose: number analyzed (Participants) | 52 | 51
  1 hours Post-dose | 3.4 [1.14 to 5.69] | -2.0 [-4.29 to 0.27]
  2.5 hours Post-dose | 6.2 [4.28 to 8.16] | -2.3 [-4.27 to -0.38]
  4 hours Post-dose | 7.5 [5.54 to 9.44] | -1.1 [-3.06 to 0.84]
  8 hours Post-dose | -1.3 [-3.53 to 0.86] | -9.9 [-12.05 to -7.66]
  12 hours Post-dose | 0.1 [-2.16 to 2.27] | -6.8 [-9.05 to -4.61]
  24 hours Post-dose: number analyzed (Participants) | 51 | 52
  24 hours Post-dose | 3.9 [2.14 to 5.75] | -2.2 [-3.97 to -0.37]
Statistical Analysis 1: Comparison: Moxifloxacin vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QTcF (ms) at 0.5 Hours Post-dose; LS Mean = 1.2, 90% CI 2-sided [-1.64 to 4.04], Standard Error of Mean 1.71
Statistical Analysis 2: Comparison: Moxifloxacin vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QTcF (ms) at 1 Hours Post-dose; LS Mean = 5.4, 90% CI 2-sided [2.22 to 8.63], Standard Error of Mean 1.93
Statistical Analysis 3: Comparison: Moxifloxacin vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QTcF (ms) at 2.5 Hours Post-dose; LS Mean = 8.5, 90% CI 2-sided [5.81 to 11.28], Standard Error of Mean 1.64
Statistical Analysis 4: Comparison: Moxifloxacin vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QTcF (ms) at 4 Hours Post-dose; LS Mean = 8.6, 90% CI 2-sided [5.86 to 11.34], Standard Error of Mean 1.65
Statistical Analysis 5: Comparison: Moxifloxacin vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QTcF (ms) at 8 Hours Post-dose; LS Mean = 8.5, 90% CI 2-sided [5.43 to 11.61], Standard Error of Mean 1.86
Statistical Analysis 6: Comparison: Moxifloxacin vs Placebo; Test type: Other — Placebo-corrected change-from-baseline QTcF (ms) at 12 Hours Post-dose; LS Mean = 6.9, 90% CI 2-sided [3.76 to 10.00], Standard Error of Mean 1.88
Statistical Analysis 7: Comparison: Moxifloxacin; Test type: Other — Placebo-corrected change-from-baseline QTcF (ms) at 24 Hours Post-dose; LS Mean = 6.1, 90% CI 2-sided [3.58 to 8.62], Standard Error of Mean 1.52

29. Secondary Outcome: Percentage of Participants With Treatment Emergent Adverse Events
Time Frame: Up to approximately 20 weeks.
Population: Groups C&D together are positive control to balovaptan. Moxifloxacin is given in a nested cross-over way using a joint placebo/positive control period, half subjects dosed with moxifloxacin on Day 2 and other half dosed on Day 15.
Measure: Number; unit: Percentage of Participants
Arm/Group | Treatment Sequence A and B and Either C or D
Number analyzed (Participants) | 57
Percentage of Participants | 42.1

ADVERSE EVENTS:
Time Frame: From the first study drug to the data cutoff date: 13 July 2019 (up to 20 weeks)
Groups:
- Treatment A Dose Level A: Participants in treatment A received balovaptan at dose level A.
- Treatment B Dose Level B: Participants in treatment B received balovaptan at dose level B.
- Treatment C Placebo + Moxifloxacin 400 mg Day 2: Participants in treatment C received placebo plus 400 mg of moxifloxacin on Day 2.
- Treatment D Placebo + Moxifloxacin 400 mg Day 15: Participants in treatment D received placebo plus 400 mg moxifloxacin on Day 15.
- All Participants: All participants received Treatment A and Treatment B and either Treatment C or Treatment D.
Arm/Group | Treatment A Dose Level A | Treatment B Dose Level B | Treatment C Placebo + Moxifloxacin 400 mg Day 2 | Treatment D Placebo + Moxifloxacin 400 mg Day 15 | All Participants
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/52 | 0/26 | 0/26 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/52 | 0/26 | 0/26 | 0/57
Other Adverse Events (participants affected / at risk) | 11/55 | 3/52 | 6/26 | 5/26 | 18/57
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A Dose Level A (N=55) | Treatment B Dose Level B (N=52) | Treatment C Placebo + Moxifloxacin 400 mg Day 2 (N=26) | Treatment D Placebo + Moxifloxacin 400 mg Day 15 (N=26) | All Participants (N=57)
Headache (Nervous system disorders) | 9 | 3 | 5 | 4 | 15
Constipation (Gastrointestinal disorders) | 3 | 0 | 1 | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-04-23): https://cdn.clinicaltrials.gov/large-docs/98/NCT03808298/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-07): https://cdn.clinicaltrials.gov/large-docs/98/NCT03808298/SAP_001.pdf